CLINICAL TRIAL: NCT01248195
Title: Optimization of Treatment and Management of Schizophrenia in Europe
Acronym: OPTIMISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rene Kahn (Other)
Collaborators: King's College London (Other); Technical University of Munich (Other); University of Manchester (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor-Investigator, Rene Kahn, MD PhD, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KP7242114; 2010-020185-19 (EudraCT Number)
Record Dates: First submitted 2010-10-20; First posted 2010-11-25 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorder
Keywords: Schizophrenia; Schizophreniform disorder; Schizoaffective disorder; Imaging; Prognosis; Treatment guidelines; Pharmacogenetics
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Phase I: 1 arm 'amisulpride open label' (Other): For 4 weeks, all patients will be treated with amisulpride open label.
  Interventions: Drug: Amisulpride open label
- Phase II: 'amisulpride double blind' (Active Comparator): Patients who do not meet remission criteria during phase I (4 weeks open label amisulpride), flow to phase II where they are randomised to 1 of 2 6-week double blind treatment arms, one of which is 'amisulpride double blind'
  Interventions: Drug: 6-week amisulpride double blind treatment
- Phase II 'olanzapine double blind' (Active Comparator): Patients who do not meet remission criteria during phase I (4 weeks open label amisulpride), flow to phase II where they are randomised to 1 of 2 6-week double blind treatment arms, one of which is 'olanzapine double blind'
  Interventions: Drug: 6-week olanzapine double blind treatment
- Phase III: 1 arm 'clozapine open label' (Other): Patients who do not meet remission criteria during phase II (6-week double blind amisulpride vs olanzapine), flow to phase III, where only 1 arm is available: 'clozapine open label'
  Interventions: Drug: 12-week clozapine open-label treatment
- Psychosocial intervention (Experimental): Patients who meet remission criteria during any of the phases of the medication component, patients who drop out of the medication component and patients who did not meet remission criteria at the end of the medication component, will flow to the psychosocial intervention component, where they are randomised to 1 of 2 arms, one of which is the 'Psychosocial Intervention' arm.
  Interventions: Behavioral: Psychosocial intervention
- Psychosocial Intervention phase: 'TAU' (No Intervention): Patients who meet remission criteria during any of the phases of the medication component, patients who drop out of the medication component and patients who did not meet remission criteria at the end of the medication component, will flow to the psychosocial intervention component, where they are randomised to 1 of 2 arms, one of which is the 'Treatment as usual' arm.

INTERVENTIONS:
Drug: Amisulpride open label — 4-week open label amisulpride treatment
  Arms: Phase I: 1 arm 'amisulpride open label'
Drug: 6-week amisulpride double blind treatment — 6-week amisulpride double blind treatment
  Arms: Phase II: 'amisulpride double blind'
Drug: 6-week olanzapine double blind treatment — 6-week olanzapine double blind treatment
  Arms: Phase II 'olanzapine double blind'
Drug: 12-week clozapine open-label treatment — 12-week clozapine open-label treatment
  Arms: Phase III: 1 arm 'clozapine open label'
Behavioral: Psychosocial intervention — Psychosocial intervention
  Arms: Psychosocial intervention

SUMMARY:
The purpose of the study is optimising current treatments in schizophrenia and explore novel therapeutic options for schizophrenia. The study intends to both address basic, but so far unanswered, questions in the treatment of schizophrenia and develop new interventions. It is expected that the project will lead to evidence that is directly applicable to treatment guidelines, and will identify potential mechanisms for new drug development.

DETAILED DESCRIPTION:
Despite nearly fifty years of pharmacological and psychosocial research, the overall prognosis of schizophrenia has improved only marginally. While the efficacy of most antipsychotic medication is generally uncontested, their overall functional impact has been modest. In order to improve this unsatisfactory result, this study aims to optimize current treatments in schizophrenia and explore novel therapeutic options for schizophrenia. The study comprises a medication intervention component, a psychosocial intervention component, a biological predictor component and an MRI component. MRI assessments are performed at baseline, and used to determine whether potential organic causes for psychotic symptoms are present, and to test prospective value of these assessments for subsequent treatment response. MRI assessments of healthy volunteers will be included to test for deviations in patients' assessments; these volunteers will not participate in any other protocol procedure. The medication intervention component comprises a first 4-week phase of amisulpride treatment. Non-responders will subsequently be randomised to a 6-week double blind phase on either amisulpride or olanzapine. Patients who classify as non-responders at the end of this phase, a 12-week open label treatment with clozapine is initiated. Patients who classify as a responder in phase I, II or III, are drop outs or who are non-responders at the end of phase III flow to the psychosocial intervention component of the study. During this part, several interventions are tested, aimed to increase treatment compliance and keep patients on the medication to which they've responded well. Through the biological predictor component, it is determined whether glutamatergic markers predict response to first and second line treatments, and if an empirical combination of pharmacogenetic, proteomics- and metabolomic markers can provide clinical valuable predictive value.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia as defined by DSM-IV-R as determined by the M.I.N.I.plus
2. Age 18 or older.
3. The first psychosis occurred at least one year and no more than 7 years ago.*
4. If patients are using an antipsychotic drug, a medication switch is currently under consideration.
5. Capable of providing written informed consent.

Exclusion Criteria:

1. Intolerance / hypersensitivity to one of the drugs (including active substances, metabolites and excipients) in this study including oral risperidone, paliperidone and aripiprazole and/or hypersensitivity to risperidone.
2. Pregnancy or lactation.
3. Patients who are currently using clozapine.
4. Patients who do not fully comprehend the purpose or are not competent to make a rational decision whether or not to participate.
5. Patients with a documented history of non-response and/or intolerance to any of the study medications and/or a documented history of non-response to a treatment with one of the study drugs of at least 6 weeks within the registered dose range.
6. Forensic patients.
7. Patients who have been treated with an investigational drug within 30 days prior to screening.
8. Simultaneous participation in another intervention study (neither medication or psychosocial intervention).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 479 (Actual)
Dates: Start 2011-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
PANSS | Jan 2016
  Study consists of multiple components, each with their own objectives. For this (medication) component: number of patients in remission, based on PANSS scores (criteria of Andreasen et al.; 2005) after 4 weeks open label amisulpride, after 6 weeks double blind amisulpride or olanzapine and after 12 weeks of open label clozapine.
Sellwood rating scale | Jan 2016
  Psychosocial intervention component, objective A: drug adherence rates as a function of (standardized self report and) Sellwood rating scales after 12 and 52 weeks.
Biological profile | jan 2016
  Biological predictors component, objective A: drug response (remission vs non-remission) as a function of biological profile, after 4 weeks, 10 weeks and 22 weeks (after each medication phase).
MRS measures | jan 2016
  Biological predictors component, objective B: using MRS scans, differences between responders and non-responders in regional glutamate levels a) at baseline and b) between baseline and after one month of treatment with amisulpiride.
SOFAS global functioning | jan 2016
  Psychosocial intervention component, objective B: drug adherence rates as a function of standardized global functioning (SOFAS score after 1 year) following psychosocial intervention vs treatment as usual.
MRI assessments | jan 2016
  MRI component objective: the percentage of first episode patients that show radiological abnormalities suggestive of neurological disorders which may explain the occurrence of psychotic symptoms - measurement at baseline only.

SECONDARY OUTCOMES:
All cause treatment discontinuation | jan 2016
  The different components of the study have their own secondary objectives:
  Medication component has multiple secondary objectives, most important one is all-cause treatment discontinuation after 4 weeks, 10 weeks and 22 weeks. Number and reason for premature discontinuations (treatment discontinuation) of the amisulpride and the olanzapine group will be compared (after 10 weeks).
All cause discontinuation | jan 2016
  Psychosocial intervention component has multiple secondary objectives, most important one is all-cause treatment discontinuation between treatment groups after 12 and 52 weeks.
Biological markers | jan 2016
  Biological predictors component has multiple secondary objectives, most important one is the ability of biological markers to predict response to antipsychotic and treatment tolerability in schizophrenia, after 4, 10 and 22 weeks.
MRI assessments | jan 2016
  The ability of MRI to predict response to antipsychotic treatment in schizophrenia, after 4, 10 and 22 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: René Kahn, MD, PhD, Principal Investigator — University Medical Center Utrecht, the Netherlands
Locations (26):
- Melbourne Neuropsychiatry Centre, Melbourne, Australia
- Department of Biological Psychiatry, Innsbruck University Clinics, Innsbruck, Austria
- Katholieke Universiteit Leuven (KU Leuven), Leuven, Belgium
- University Specialised Hospital for Active Treatment in Neurology and Psychiatry "St. Naum", Sofia, Bulgaria
- Czechia (2):
  - Psychiatrické centrum Praha, Prague, Ustavni 91
  - Psychiatrická klinika LF UK, Fakultní nemocnice, Hradec Králové
- Center for Neuropsychiatric Research, Glostrup Municipality, Denmark
- Institut National de la Santé et de la Reserche Médicale (INSERM), Créteil, France
- Germany (4):
  - Martin-Luther-University (MLU) of Halle-Wittenberg, Halle
  - Deprtment of Psychiatry, University of Heidelberg, Mannheim
  - Ludwig-Maximilians University München, München
  - Technische Universität München (TUM), München
- Sheba Medical Centre Department of Psychiatry, Tel Litwinsky, Israel
- Department of Psychiatry University of Naples, Naples, Italy
- University Medical Center Utrecht, Utrecht, Netherlands
- Department of Adult Psychiatry, University of Medical Sciences, Poznan, Poland
- Obregia Psychiatric Hospital, Bucharest, Romania
- Spain (5):
  - Hospital Clinic i Provincial, Barcelona
  - Servicio Madrileño de Salud (SERMAS), Madrid
  - Hospital Clínico San Carlos, Madrid
  - Instituto de Investigación Hospital 12 de Octubre, Madrid
  - Universidad de Oviedo, Oviedo
- Clienia Schlössli AG, Privatklinik für Psychiatrie und Psychotherapie, Oetwil, Switzerland
- United Kingdom (3):
  - King's College London, Departments of Psychological Medicine, Psychiatry & Cognitive Neuroscience, London
  - West London Mental Health Trust, London
  - University of Manchester, Manchester

REFERENCES:
- [Derived] Nasib LG, Winter-van Rossum I, Zuithoff NPA, Boudewijns ZSRM, Leucht S, Kahn RS. Generalizability of the Results of Efficacy Trials in First-Episode Schizophrenia: Comparing Outcome and Study Discontinuation of Groups of Participants in the Optimization of Treatment and Management of Schizophrenia in Europe (OPTiMiSE) Trial. J Clin Psychiatry. 2023 Mar 29;84(3):22m14531. doi: 10.4088/JCP.22m14531. PMID 36988483
- [Derived] Fraguas D, Diaz-Caneja CM, Pina-Camacho L, Winter van Rossum I, Baandrup L, Sommer IE, Glenthoj B, Kahn RS, Leucht S, Arango C. The role of depression in the prediction of a "late" remission in first-episode psychosis: An analysis of the OPTiMiSE study. Schizophr Res. 2021 May;231:100-107. doi: 10.1016/j.schres.2021.03.010. Epub 2021 Apr 7. PMID 33838518
- [Derived] Pollak TA, Vincent A, Iyegbe C, Coutinho E, Jacobson L, Rujescu D, Stone J, Jezequel J, Rogemond V, Jamain S, Groc L, David A, Egerton A, Kahn RS, Honnorat J, Dazzan P, Leboyer M, McGuire P. Relationship Between Serum NMDA Receptor Antibodies and Response to Antipsychotic Treatment in First-Episode Psychosis. Biol Psychiatry. 2021 Jul 1;90(1):9-15. doi: 10.1016/j.biopsych.2020.11.014. Epub 2020 Nov 24. PMID 33536130
- [Derived] Kahn RS, Winter van Rossum I, Leucht S, McGuire P, Lewis SW, Leboyer M, Arango C, Dazzan P, Drake R, Heres S, Diaz-Caneja CM, Rujescu D, Weiser M, Galderisi S, Glenthoj B, Eijkemans MJC, Fleischhacker WW, Kapur S, Sommer IE; OPTiMiSE study group. Amisulpride and olanzapine followed by open-label treatment with clozapine in first-episode schizophrenia and schizophreniform disorder (OPTiMiSE): a three-phase switching study. Lancet Psychiatry. 2018 Oct;5(10):797-807. doi: 10.1016/S2215-0366(18)30252-9. Epub 2018 Aug 13. PMID 30115598